CLINICAL TRIAL: NCT04174794
Title: Investigating Reduction of aCute heArt Failure Readmission With Lung UltraSound-preliminary Trial (Pre-IcarUS)
Brief Title: Investigating Reduction of aCute heArt Failure Readmission With Lung UltraSound-preliminary Trial
Acronym: Pre-IcarUS
Status: Terminated | Type: Observational
Why Stopped: COVID-19 Pandemic
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Antonio Leidi, Principal Investigator, University Hospital, Geneva
Other Study IDs: 2019-01596
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Acute Heart Failure
Keywords: Acute heart failure; Lung ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Lung ultrasound — The two different lung ultrasound protocols are performed initially within 48 hours of internal medicine ward admission by a pair of expert-beginner echographers. In case of admission during non-working days, the first scan can be done within 72 hours from admission. Follow-up scans are repeated 4 to 6 days later or on the day of discharge if it occurs before de fourth day. Experts and beginners execute the lund ultrasound protocols in sequence, reciprocally blinded, without accessing to clinical data files.
  Other Names: Philips Sparq® ultrasound system; Philips AG Health Systems

SUMMARY:
In Switzerland 15% of discharged patients are readmitted within 30 days. Acute heart failure is the leading cause of hospital admission and one of the most frequent reasons for re-admission, mainly because of congestion-driven symptoms. Residual congestion is noted in 10%-15% of patients at discharge and is associated with an increased risk of re-admission and mortality. Lung ultrasound outperforms both chest X-ray and physical examination in detection of lung congestion. Several semiquantitative scanning protocols exist for quantifying congestion. The aim of this study is to compare for the first time two widely used lung ultrasound protocols, one exhaustive (28-points) and one simplified (8-points), in real-time settings. The focus is placed on reproducibility (expert-beginner interobserver concordance), feasibility (time consumption for images acquisition and interpretation) and performance (detection of B-lines clearing) of both scores. Semi-quantitative method is expected to have better feasibility with similar reproducibility and performance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute heart failure on admission chart (primary or secondary diagnosis)
* Admission from the emergency room to a general internal medicine ward
* Presentation of acute heart failure according to European Society of Cardiology :
* Presence of ≥1 symptom or sign based on admission chart review and
* Raised value of N terminal-pro-brain natriuretic peptide (>300 ng/l)

Exclusion Criteria:

* Interstitial lung disease, lung cancer or metastasis, acute respiratory distress syndrome, pulmonary contusion, previous lung surgery
* Inability or unwillingness to give consent
* Presence of oligo-anuric end stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A convenience sample of 90 patients admitted to from the emergency room to a general internal medicine ward of a tertiary care center with the diagnosis of acute heart failure
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Inter-observer disagreement at admission lung ultrasound | Day 0
  The primary endpoint is the amount of disagreement between beginner and expert echographers at admission lung ultrasound. In order to compare protocols using different grading systems, a common 4-levels interstitial syndrome (IS) severity scale is defined. For the 28-point protocol, rating of total number of B-lines will be classified according to literature in severe (>30), moderate (16-30), mild (6-15) or no signs of IS (≤5 B-lines). For the 8-point protocol, IS is arbitrarily classified as follows: 'severe' (6-8), 'moderate' (4-5), mild (2-3) and 'no signs' (0-1 positive zones).
Inter-observer disagreement at follow-up lung ultrasound | Day 4 to 6
  The amount of disagreement between beginner and expert echographers is measured at follow-up lung ultrasound. In order to compare protocols using different grading systems, a common 4-levels IS severity scale is defined. For the 28-point protocol, rating of total number of B-lines will be classified according to literature in severe (>30), moderate (16-30), mild (6-15) or no signs of IS (≤5 B-lines). For the 8-point protocol, IS is arbitrarily classified as follows: 'severe' (6-8), 'moderate' (4-5), mild (2-3) and 'no signs' (0-1 positive zones).

SECONDARY OUTCOMES:
Time consumption for images acquisition and interpretation at admission lung ultrasound | Day 0
  The time spent for images acquisition and interpretation is measured in both 28-point and 8-point protocols.
Time consumption for images acquisition and interpretation at follow-up lung ultrasound | Day 4 to 6
  The time spent for images acquisition and interpretation is measured in both 28-point and 8-point protocols.
Change in interstitial syndrome severity scale and amount of B-lines at follow-up ultrasound from baseline | Day 0, Day 4 to 6
  The clearing of B-lines following decongestive therapy is analysed and correlated to a clinical congestion score evolution, the loss of weight, N terminal-pro-brain natriuretic peptide value decline.
Post-discharge readmission and mortality at 30 days | Day 30 post-discharge
  The analysis of correlation between admission, follow-up lung ultrasound IS, echographic decongestion (i.e. B-lines clearing) with readmission and mortality at 30 days post-discharge
Post-discharge readmission and mortality at 60 days | Day 60 post-discharge
  The analysis of correlation between admission, follow-up lung ultrasound IS, echographic decongestion (i.e. B-lines clearing) with readmission and mortality at 60 days post-discharge
Post-discharge readmission and mortality at 90 days | Day 90 post-discharge
  The analysis of correlation between admission, follow-up LUS ISSS, echographic decongestion (i.e. B-lines clearing) with readmission and mortality at 90 days post-discharge
Post-discharge readmission and mortality at 180 days | Day 180 post-discharge
  The analysis of correlation between admission, follow-up lung ultrasound IS, echographic decongestion (i.e. B-lines clearing) with readmission and mortality at 180 days post-discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No